CLINICAL TRIAL: NCT01569893
Title: RENEWING HEALTH - Large Scale Pilot in Veneto Region: Life-long Monitoring of Diabetes Mellitus
Brief Title: Life-Long Monitoring of Diabetes Mellitus in Veneto Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regione Veneto (Other)
Collaborators: European Commission (Other); Azienda ULSS 4 Alto Vicentino (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: G. A. 250487 - Veneto WP8Cl2
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2014-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Telemonitoring; Telemedicine; Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Usual care: treatment as usual
- Self-monitoring for patients with Dibetes mellitus type 2 (Experimental): Self-monitoring for patients with Dibetes mellitus type 2
  Interventions: Other: Self-monitoring for patients with Dibetes mellitus

INTERVENTIONS:
Other: Self-monitoring for patients with Dibetes mellitus — Patients are equipped with a telemonitoring kit composed by a portable glucose meter and a gateway device for data transmission.
  The patient can monitor his blood glucose level with a frequency set by the clinician in the personalised treatment plan. Data are transmitted to a regional eHealth centre where a group of operators keeps these information under control and alert the reference clinician in case of worsening of symptoms.
  Arms: Self-monitoring for patients with Dibetes mellitus type 2

SUMMARY:
To evaluate whether patients with type 2 diabetes mellitus can be followed by simplified, centralized and large scale tele-monitoring of blood glucose levels, and whether this intervention produces health and economic benefits when introduced without major changes to the existing organization of a large treatment care center.

DETAILED DESCRIPTION:
The study is designed to evaluate the impact of telemonitoring on the management of Diabetes Mellitus compared with outpatient usual care. From a clinical point of view, the measurements of HbA1c will be taken to assess glycaemic control and the trial will allow to investigate how telemonitoring contributes to improve Diabetes mellitus patients health-related quality of life and reduct the access to hospital facilities (re-hospitalizations, bed-days, specialistic and ER visits) and the anxiety about health conditions. A cost-effectiveness and cost-utility analysis will be carried out in order to determine if and how telemonitoring helps to limit the healthcare expenditure. The evaluation will deal also with organizational changes and task shift due to telemonitoring introduction and patients and professionals perception towards the service.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 Diabetes
* HbA1c > 53 mmol/mol (7.0 % according to NGSP)
* Capability to use the devices provided
* Being cognitively able to participate
* Capability of filling in questionnaires in german or greek or italian language
* Absence of severe comorbidity prevalent on diabetes with life expectancy < 12 months

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Health related quality of life of the patients measured by the SF-36 version 2 questionnaire | At the entry point of intervention and at the end (12 months)
Glycated hemoglobin (HbA1c) levels | At the entry point of intervention and at the end (12 months)

SECONDARY OUTCOMES:
Number of hospitalisations. | 12 months
Number of hospitalisations due to diabetes. | 12 months
Bed days of care | 12 months
Bed days of care due to diabetes. | 12 months
Number of visits with specialists | 12 months
Number of access to ER | 12 months
Mental status measured through Hospital Anxiety and Depression Scale (HADS). | At the entry point of intervention and at the end (12 months)
Number of visits with specialists in diabetic center | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Calcaterra, MD, Principal Investigator — Local Health Authority "Alto Vicentino" of Thiene (VI)
Locations (1):
- "De Lellis" Hospital - Diabetology-Endocrinology Department, Schio, Vicenza, Italy

REFERENCES:
- See also: Related Info — http://www.renewinghealth.eu